CLINICAL TRIAL: NCT05493553
Title: Effects of an Intermittent Fasting and Dietary Supplement Regimen on Glycemic Variability and Glycemic Control in Men and Women With Risk Factors for Impaired Fasting Glucose: A Sub-chronic Continuous Glucose Monitoring Pilot Study
Brief Title: Effects of an Intermittent Fasting and Dietary Supplement Regimen on Glycemic Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unicity International, Inc. (Industry)
Collaborators: Biofortis Innovation Services (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: BIO-2206
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Healthy; Impaired Glucose Tolerance
Keywords: Intermittent fasting; Yerba mate; Continuous glucose monitoring; Dietary supplements; Soluble fiber
MeSH Terms: conditions — Glucose Intolerance; Intermittent Fasting | interventions — diisopropyl sebacate; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Baseline (no supplements or intermittent fasting requirements) and two interventional phases (Phase 1: supplements only; Phase 2: supplements and intermittent fasting)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline (No Intervention): A baseline period (no supplements or intermittent fasting).
- Phase 1 (Experimental): A four-day period during which subjects will take a yerba mate supplement once per day in the morning and a fiber-based supplement twice per day prior to two meals.
  Interventions: Dietary Supplement: Dietary supplement regimen
- Phase 2 (Experimental): A four-day period during which subjects will take a yerba mate supplement once per day in the morning and a fiber-based supplement twice per day prior to two meals, while also practicing daily intermittent fasting (16 hours fasting, 8 hours eating window).
  Interventions: Other: Dietary supplement and intermittent fasting regimen

INTERVENTIONS:
Dietary Supplement: Dietary supplement regimen — The powdered, soluble fiber-based supplement contains soluble fibers, phytosterols, plant-derived polysaccharides, flavor, maltodextrin, orange juice powder, citric acid, vitamin and mineral blend, and sweetener. This is prepared in water and consumed twice per day, prior to a meal.
  The yerba mate-based supplement (containing green yerba mate leaf extract, sweeteners, and flavor) is a powdered supplement prepared in water and consumed in the morning.
  Other Names: Balance; Unimate
  Arms: Phase 1
Other: Dietary supplement and intermittent fasting regimen — The dietary supplement regimen is the same as in Phase 1. The intermittent fasting protocol consists of a 16-hour fasting period and an 8-hour eating window.
  Other Names: Feel Great
  Arms: Phase 2

SUMMARY:
The purpose of this study is to determine the short-term effect of a nutritional program consisting of a yerba mate supplement, fiber supplement, and intermittent fasting on glycemic variability in men and women with risk factors for impaired fasting glucose.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of a nutritional program which combines two different supplements (a yerba mate extract supplement and a fiber-based, vitamin-rich nutritional supplement) and intermittent fasting on glycemic variability and glycemic control in men and women with risk factors for impaired fasting glucose.

This study will be an exploratory pilot study with one screening visit, one baseline visit followed by a baseline phase, two intervention phases, and one follow-up visit. During the baseline phase, subjects will follow their regular dietary routines. During the 4-day Phase 1, subjects will take the yerba mate supplement once per day and the fiber supplement twice per day. During the 4-day Phase 2, subjects will continue the supplement regimen from Phase 1, while incorporating daily intermittent fasting for approximately 16 hours and eating for 8 hours. A continuous glucose monitor will be worn by each subject to continuously measure glucose throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥25.0 to <35.0 kg/m2

At least 1 out of the 3 following criteria:

* Waist circumference >102 cm for men and >88 cm for women
* Family history of at least one parent or sibling with diagnosed impaired fasting glucose (IFG) or type 2 diabetes mellitus (T2DM)
* Sedentary lifestyle (based on self-report)

Exclusion Criteria:

* Fasting glucose ≥126 mg/dL or diagnosed with diabetes mellitus (type 1 or 2).
* Uncontrolled and/or clinically important pulmonary, hepatic, renal, cardiac, hematologic, immunologic, neurologic, psychiatric or biliary condition(s). Conditions which are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
* Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg)
* History of or current diagnosis of conditions that may affect blood glucose levels.
* Any known food allergy as well as intolerance or sensitivity to study product ingredients and caffeine.
* Any extreme diets or history of eating disorders that in the opinion of the Clinical Investigator that may affect the study outcomes or the subject's ability to adhere to the study program.
* Weight loss or gain > 4.5 kg within 90 days of Visit 1.
* Currently or planning to be on a weight loss or weight gain / muscle-building regimen program during the study.
* Major trauma or any other surgical event within 90 days of Visit 1.
* History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Unstable use of hormonal contraceptives (change in medication regimen within 90 days of Visit 1).
* Unstable use of medications that affect blood glucose levels whereby stable is defined as no change in regimen within 90 days of Visit 1.
* Use of oral or injectable steroids (topical and inhaled are allowed) within 90 days of Visit 1
* Use of fiber supplements or intentionally increasing fiber intake within 30 days of Visit 1
* Use of yerba mate containing products (beverage, supplement) within 30 days of Visit 1
* Exposure to any non-registered drug product within 30 days prior to Visit 1
* Use of vitamin C-containing supplements (including multivitamins) within 24 hours of Visit 2 and during the study intervention period.
* Use of products containing salicylic acid (skin-care products are allowed if not used on the area surrounding the sensor) within 24 hours of Visit 2 and during the study intervention period.
* Use of topical marijuana or hemp products within 24 hours of Visit 2 and during the study intervention period.
* Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception during the study period.
* Recent history (within 12 months) of alcohol or substance abuse.
* Has a condition the Clinical Investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Glycemic variability | 3 days
  Within-subject change in glucose coefficient of variation (CV)

SECONDARY OUTCOMES:
Daytime and Overall Blood Glucose Levels | 3 days
  Daytime (6 am - 11:59 pm), Overall (24 hours)
Daytime glycemic variability | 3 days
  Coefficient of variation (CV) of glucose values during daytime hours (6 am - 11:59 pm)
Percent of time in range | 3 days
  70-140 mg/dL
Percent of time below range | 3 days
  < 70 mg/dL
Percent of time above range | 3 days
  > 140 mg/dL
Gastrointestinal symptoms | 2 weeks
  Daily gastrointestinal tolerance questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Beckman, MD, Principal Investigator — Biofortis Innovation Services
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States